CLINICAL TRIAL: NCT07387601
Title: Effect of Peer-led Educational Intervention on Treatment Outcomes Among Adults With Drug-susceptible Pulmonary Tuberculosis in South Omo and Ari Zone, Southern Ethiopia: A Protocol for a Cluster- Randomized Controlled Trial Study
Brief Title: Effect of Peer-led Educational Intervention on Treatment Outcomes Among Adults With Drug-susceptible Pulmonary Tuberculosis in South Omo and Ari Zone, Southern Ethiopia
Acronym: DS-PTB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahirdar University (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4064/2024
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: to Assess Effect of Peer-led Education
Keywords: Southern Ethiopia south omo

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial with a parallel assignment design to evaluate the effect of a peer-led educational intervention on treatment outcomes, quality of life, disability, and depression among adult tuberculosis patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- peer-led educational intervention (Active Comparator): The intervention includes health education, behavioral counseling, skills training, and supportive follow-up aimed at reducing depressive symptoms, disability level and improving quality of life and Treatment successes rate among TB patients
  Interventions: Combination Product: peer-led education

INTERVENTIONS:
Combination Product: peer-led education — The Intervention is a structured, evidence-based program designed to promote positive and sustained behavioral changes among participants through education, counseling, and supportive follow-up

SUMMARY:
The study might come up with valuable findings to address poor treatment outcome, poor quality of life, disability score and depressive symptoms. The findings may also be decreased health professional workload. The findings would be supportive evidences for policy makers, program managers, to clinician as well as the patients themselves and for other researchers. The study may help to promote and maintain good treatment outcome for the patients in the study area as well as the country. The findings will also be used for teaching & learning purposes in educational & training programs.

DETAILED DESCRIPTION:
Peer-led education is an effective approach in improving knowledge and attitude. It is also helpful to reach specific marginalized populations, to reduce social stigma and to enhance adherence by improving behavioral outcomes since behaviour is socially influenced and behavioral norms are developed through social interaction. Peers are underused resources for strengthening TB control and prevention because they have a unique power to support socially excluded patients through sharing their personal experience, to affirm previous beliefs and intentions, and to inspire future opportunities. Peers are more preferred than TB focal persons because they act as a friend, as an educator, as an activist, as a role model and as a team member but TB focal persons act only as an educator. So, this manual is organized to improve knowledge and attitude towards tuberculosis, to reduce social stigma and to strengthen TB control and prevention strategies

ELIGIBILITY:
Inclusion Criteria:

* Adults with new drug-susceptible pulmonary TB who will be diagnosed in bacteriological diagnostic methods
* not participating in similar study,
* mentally capable to provide consent,
* physically capable of following the intervention.

Exclusion Criteria:

* Seriously ill patients at the time of screening or enrollment
* Tuberculosis patients with a known plan to be transferred out of the study sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-07-12 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
treatment success rate | the primary outcome will be measured at the end of 6 months i.e after July 24/2026
  as defined by 7th edition of Ethiopian guidelines for clinical and programmatic management of TB, TB/HIV, DR-TB and Leprosy and by WHO. Data on the patients' status on the primary outcome variable will be extracted from TB register logbook.

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data (IPD) will be shared: demographic information (age, sex, ethnicity), clinical measurements (blood pressure, weight, laboratory test results), questionnaire responses (PHQ-9 scores for depression, quality of life scores), and study outcomes (treatment response, adverse events). All data will be de-identified to protect participant privacy
Supporting Information: Study Protocol
Time Frame: February 10/2026-July 24/2026
Access Criteria: up on the request the correspondence author
URL: https://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration

REFERENCES:
- [Result] Authors (full names or at least last name + initials, in order) Article title Journal name Publication date (year, and month if available) Volume number Page numbers